CLINICAL TRIAL: NCT00682721
Title: Valacyclovir Suppression to Improve the Stability of Vaginal Flora Among HSV-2 Seropositive Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor has withdrawn support for this study and it will not be performed
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Thomas L. Cherpes, MD, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO 08090230
Record Dates: First submitted 2008-05-16; First posted 2008-05-22 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Bacterial Vaginosis; Herpes Simplex Virus Type II
Keywords: Bacterial Vaginosis; Herpes Simplex Virus Type II
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Valacyclovir 1 gm daily x number of days active in the study
  Interventions: Drug: Valacyclovir
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Matching placebo two pills once daily
  Arms: 1
Drug: Valacyclovir — 1 gram daily x number of days active in the study
  Arms: 2

SUMMARY:
We will be examining the effects of suppressive valacyclovir therapy on the stability of vaginal flora in women who are seropositive for HSV-2. We have preliminary data that suggests the presence of HSV-2 increases the risk for Group B Streptococcus colonization as well as many other deleterious organisms (e.g. Streptococcus pseudoporcinus), in addition to increasing the risk for acquisition of BV-associated vaginal flora. We will be examining the effects of suppressive therapy on the vaginal flora of any HSV-2 seropositive woman.

ELIGIBILITY:
Screening Inclusion Criteria:

* Women 18-40 years of age at the time of screening
* Willing to be screened for HSV-2 using a rapid, FDA approved test
* Using an effective method of birth control (examples of effective methods of birth control are: women practicing abstinence x 90 days, hormonal birth control, consistent condom use, bilateral tubal ligation, partner with a vasectomy)

Screening Exclusion Criteria:

* Pregnant or nursing mother
* Use of any antimicrobial agents (vaginal or systemic) for the treatment of any condition within 7 days
* Presence of any intrauterine device
* Allergy or hypersensitivity to valcyclovir or nucleoside analogues

Enrollment Inclusion Criteria:

* Women 18-40 Years of age at the time of screening
* HSV-2 seropositive as determined by rapid HSV-2 testing
* Using an effective method of birth control (examples of effective methods of birth control are: women practicing abstinence x 90 days, hormonal birth control, consistent condom use, bilateral tubal ligation, partner with a vasectomy)
* Willing to avoid use of any intravaginal products during study period
* Capable of providing written informed consent
* Capable of cooperating to the extent and degree required by this protocol

Enrollment Exclusion Criteria:

* Pregnancy (all women will have a urine pregnancy test prior to randomization and treatment)
* nursing mother
* Menopausal women
* Use of any antimicrobial agents (vaginal or systemic) for the treatment of any condition within 7 days of study enrollment
* Known immunocompromised state
* Significant Medical disorder that precludes accurate evaluation of participants condition
* Presence of any intrauterine device
* History of significant hepatic or renal impairment
* Sensitivity/allergy to valacyclovir or nucleoside analogues
* history of acyclovir or valacyclovir resistant HSV infection
* Participation in a study using an investigational product in the past 30 days

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study will be a determination of the ability of valacyclovir suppressive therapy to stabilize the vaginal flora. | within 90 days of enrollment

SECONDARY OUTCOMES:
The frequency of detection of HSV-2 in the lower genital tract at the follow up visits. | within 90 days of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Cherpes, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States